CLINICAL TRIAL: NCT00000212
Title: IV Cocaine Abuse: A Laboratory Model
Brief Title: IV Cocaine Abuse: A Laboratory Model - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-06234-1; R01DA006234 (NIH); R01-06234-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2012-12

CONDITIONS: Cocaine-Related Disorders
Keywords: crack cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Desipramine

INTERVENTIONS:
Drug: Desipramine

SUMMARY:
The purpose of this study is to evaluate the effects of desipramine DMI maintenance on cocaine taking and on the physiological and subjective effects of cocaine, including cocaine craving.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1987-07; Primary Completion 1988-07 (Actual); Study Completion 1988-07 (Actual)

PRIMARY OUTCOMES:
Amount cocaine self-administered
Direct cocaine effects (cardiovascular, subjective
Interaction of cocaine and DMI on cardio measures
Interaction of cocaine/DMI on coc's subjective
Effects of DMI on cocaine craving
Drug use during outpatient DMI maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Richard Foltin, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Fischman MW, Foltin RW, Nestadt G, Pearlson GD. Effects of desipramine maintenance on cocaine self-administration by humans. J Pharmacol Exp Ther. 1990 May;253(2):760-70. PMID 2338656